CLINICAL TRIAL: NCT03541096
Title: The Impact of Winter Swimming on Brown Adipose Tissue Recruitment and Metabolic Health in Middel-aged Obese Pre-diabetic Subjects.
Brief Title: Winter-Swimming and Brown Adipose Tissue Activity in Middel-aged Obese Subjects (WinterBAT).
Acronym: WinterBAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Karstoft (Other)
Responsible Party: Sponsor-Investigator, Kristian Karstoft, MD, PhD, Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-18015882 WinterBAT-Study
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-05

CONDITIONS: Adipose Tissue, Brown; Brown Adipose Tissue; Uncoupling Protein 1; Cold Exposure; Obesity; Type 2 Diabetes Mellitus; Winter Swimming
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Winter Swimmers (Experimental): 4 Months of supervised winter swimming.
  Interventions: Behavioral: Winter Swimming
- Control group (Placebo Comparator): No winter swimming activities.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Winter Swimming — Supervised Winter Swimming in Copenhagen
  Arms: Winter Swimmers
Behavioral: Control group — No winter swimming activities.
  Arms: Control group

SUMMARY:
This study investigates repetitive cold-water exposure on brown fat activity assessed by PET/CT scanning. Furthermore we will assess glucose control upon winter-swimming. Obese prediabetic men and women will be randomized to winter-swimming or control conditions for 4 months.

DETAILED DESCRIPTION:
Brown fat (BAT) is an energy-consuming tissue. Long-term activation of BAT in adults increases clearance of blood glucose and non-esterified fatty acids (NEFA), insulin sensitivity and metabolic rate. Moreover, adipokines released from BAT, known as batokines, represent a promising but currently unexplored area in terms of metabolic regulation. Cooling activates BAT; however, current cooling protocols fail to activate BAT in a large part of the population. Whether this failure in activation is related to biology, inefficient detection or cooling protocols is unknown. With our initial acute cooling study (protocol number: H-16038581), these protocols have successfully been optimized whereupon novel batokines will be identified. Having established a methodology for assessing BAT activity and batokine profiles, a longer-term cooling intervention (winter swimming) will be performed to examine the effect of repetitive cold-water exposure on BAT activity. Obese pre-diabetic subjects will be included in a 4-month supervised winter swimming (WS) intervention.

It is hypothesized, that repetitive cold-water exposure constituted by WS, increase BAT activation and volume, followed by improved glycemic control in obese pre-diabetic subjects.

Method The study is a randomized controlled, parallel-group intervention study. The investigator will recruit 30 obese pre-diabetic non-winter-swimmers to participate in a WS intervention group (n=15) or control group (n=15) with no WS activities. Subjects will either be randomized to the WS group, who will winter-swim 4 months, 2-3 times/week including sauna-visits if desired, or control conditions with no WS during the 4 months (October to May).

Main aims

* To assess whether WS will have an immediate effect on BAT recruitment or function.
* To assess whether WS will have an effect on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference above 80 cm for women and 94 cm for men.
* BMI > 25 but <40 kg/m2
* Age > 40 years.
* Low to moderate physical activity level (no physical activity or on average 30 minutes of moderate physical activity per day and not more than 3 hours of training pr. Week)

Subjects will be included in either one of these cases after the screening:

* Fasting plasma glucose above 5.6 millimol per liter (mmoL/L).
* HbA1C >39 millimol per mol (mmol/mol).
* 2 hour plasma glucose after a 75 g. oral glucose tolerance test (OGTT) above 7.8 mmol/L.

Exclusion Criteria:

* Winter swimmer
* Any history of Cancer,
* Clinically significant liver, kidney, heart, inflammatory or lung-disease.
* Pregnancy
* Taking medication (not for hay fever), including glucose-lowering treatment.
* HbA1c >55 mmol/mol and/or 2-h plasma glucose in the 75-g OGTT > 15 mmol/L, fasting plasma glucose above 6.9.
* Iron deficiency
* Increased International Normalised Ratio for coagulation (INR).
* Femoral hernia, vene prostheses (pants prosthesis), thrombs in v. Femoralis.
* Abnormal ultrasound echocardiography of the heart found at the health-examination day.
* Contraindications to cold exposure including severe Raynauds disease.
* History of alcohol abuse or use of more than 14 units pr. Week.
* History of drug abuse, including marihuana.
* Smoking including occasional smoking.
* Pacemaker or other electronics implanted in the body.
* Claustrophobia, communication problems, including understanding the experimental protocol.
* History of contrast allergy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between groups in change in brown adipose tissue (BAT) activity during cooling | Day 0 (before intervention) and Day 120 (after intervention)
  BAT activity is measured using positron emission tomography (PET)- Computer tomography (CT) scan. The PET-CT scan uses a glucose-radiotracer (fludeoxyglucose-18 (FDG)) to measure the glucose uptake in BAT, which is associated with BAT activity. FDG is injected following one hour of cooling and the subjects are scanned following one additional hour of cooling. The subjects are continuously cooled throughout the scanning procedure. Difference between groups in change in FDG tracer uptake (post minus pre intervention) during 1,5 hours of cooling is calculated.

SECONDARY OUTCOMES:
Difference between groups in change in glycemic control | Day 0 (before intervention) and Day 120 (after intervention)
  Glycemic control is measured using a 4 hour mixed meal tolerance test. Difference between groups in change in the mean MMTT glucose levels during the MMTT (post minus pre intervention) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Schéele, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Center for Inflammation and Metabolism/ Center for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No